CLINICAL TRIAL: NCT01857050
Title: Assessment of INR Prolongation in Patients Treated Simultaneously With Warfarin and Antibiotics From the Cephalosporins Family,Observational Retrospective Study.
Brief Title: Assessment of International Normalized Ratio (INR) Prolongation in Patients Treated Simultaneously With Warfarin and Cephalosporins
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC130210-12CTIL
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Many drug interactions with Warfarin are well documented in the literature, including interactions with a variety of antibiotics. However,in mamy cases it is difficult to predict when the interaction remains theoretical and when it becomes clinically significant and will be reflected in the individual patient. This study's aim is to identify and characterize related conditions (including comorbidities, laboratory test results and other parameters related to the patient)that might be predictors for drug interactions turning from theoretical to clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over
* Patients treated with a combination of Warfarin and Cephalosporins
* Patients who were hospitalized in the department of internal medicine
* Patients who were treated with Warfarin without Cefalosporins

Exclusion Criteria:

* Patients on Warfarin who did not actually receive the drug during their hospitalization
* Patients whose medical records were not accessible or didn't contain full data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Warfarin-treated patients who were hospitalized for any reason in the department of internal medicine and were treated with antibiotics from the Cephalosporins group during their hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Reasons for INR prolongation in patients who were treated with the combination of Warfarin and Cephalosporins | Participants will be followed for the duration of thei hospital stay, an expected average of 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lishner, MD, Principal Investigator — Meir Hospital, Kfar Saba, Israel